CLINICAL TRIAL: NCT00348179
Title: Vascular Function in Adolescent, Diabetic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Kurt Midyett, Children's Mercy Hospitals and Clinics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04 04-036E
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2007-04

CONDITIONS: Type 1 Diabetes
Keywords: Vascular abnormalities; Type 1 diabetes; Healthy control subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Measurement of vascular function per SphymgnoCor equipment — Pressure tonometer will be used on various vessels, non-invasive.

SUMMARY:
The objectives of this investigator initiated study are to:

1. Determine if and when vascular abnormalities occur during early adolescence
2. Determine if poor diabetic control is related to vascular abnormalities.

The development of vascular plaques and vascular contractility will be assessed through the use of the SyphmgnoCor equipment.

DETAILED DESCRIPTION:
Up to 85 Type 1 diabetic and healthy controls, 12-14 years of age, will be recruited for the study. Once the Permission/Assent form has been completed, a cuff will be applied to the arm and the pressure tonometer will be used on various vessels. Cardiovascular data will be recorded. The procedure is non-invasive, will last approximately 10 minutes and will be performed during a routine clinic visit. Onset of diabetes and level of diabetic control as measured by the most recent Hbg A1c (relative to the study visit) will be obtained from the medical record. Microalbumin levels covering the prior 12 months will be collected from the medical record of diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 12-14 years who have Type 1 diabetes or are healthy controls

Exclusion Criteria:

* Children and adolescents who do not meet inclusion criteria

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2004-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Vascular abnormalities as measured by the SyphmgnoCor equipment | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Midyett, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States